CLINICAL TRIAL: NCT04775394
Title: Activation of Apoptosis-related Receptors on Alveolar Macrophages From COPD Patients and Healthy Controls
Brief Title: Activation of Apoptosis-related Receptors on Alveolar Macrophages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jens Hohlfeld (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jens Hohlfeld, Prof. Dr. med. Jens M. Hohlfeld, Fraunhofer-Institute of Toxicology and Experimental Medicine
Organization: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20-04 ROBAL
Record Dates: First submitted 2021-02-15; First posted 2021-03-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Intervention Model Description: Enrolment will healthy subjects first, followed by subjects with COPD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Part: Healthy subjects (Experimental): 3-5 healthy ex-smokers with normal lung function to establish methods
  Interventions: Other: Bronchoscopy
- Main Part: COPD patients and Healthy Controls (Experimental): 8 subjects with COPD stage II and III who are ex-smokers and have a history of chronic cough and sputum production and 5-8 healthy, age-matched controls
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — Bronchoalveolar lavage, mucosal biopsy and bronchial brushes during bronchoscopy

SUMMARY:
The aim is to understand whether activation of receptors involved in clearance of apoptotic cells will improve efferocytosis in COPD patients in vitro and whether generation of pro-inflammatory cytokines can be decreased in COPD patients.

DETAILED DESCRIPTION:
In order to assess pathway activation in COPD macrophages, alveolar macrophages will be isolated from BAL of COPD patients and healthy controls. Alveolar macrophages will be co-cultured in vitro with apoptotic cells and treated with compounds. In addition, BAL fluid will be frozen for later testing of soluble mediators.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Able and willing to give written informed consent.
* Healthy male and female subjects, aged 18-80 years for the initial part and 40-80 years for the main part, inclusive. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs) or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
* Normal lung function with Forced Expiratory Volume in 1 second (FEV1) predicted ≥ 80% and FEV1/Forced Vital Capacity (FVC) > 70%.
* Body mass index between 18 and 32 kg/m2
* Ex-smokers since at least 12 months with a smoking history of at least 10 pack years.
* Able and willing to give written informed consent

COPD subjects

* Male and female subjects, aged 40-80 years, inclusive. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
* Clinical diagnosis of COPD stage II and III
* History of chronic cough and sputum production
* FEV1/FVC <70% post-bronchodilator at visit 1
* FEV1 30-80% of the predicted normal value post-bronchodilator at visit 1
* FEV1 >1.5 L
* Absence of lung emphysema assessed by pulmonary function measurement at visit 1: Total Lung Capacity (TLC) <120% of predicted normal, Residual Volume (RV) <120% of predicted normal, Diffusing Capacity for Carbon Monoxide (DLCO) >80%
* Ex-smokers since at least 12 months with a smoking history of at least 10 pack years.
* Body mass index between 18 and 32 kg/m2.
* Able and willing to give written informed consent.

Exclusion Criteria:

Healthy volunteers

* Past or present disease, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis)
* Regular intake of any prescribed or over the counter medication. Exceptions include paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements
* Clinically relevant history of allergy as judged by the investigator
* Intolerance against standard medication used during bronchoscopy, e.g. lidocaine, midazolam.
* Infections of the lower respiratory tract within 6 weeks prior to screening
* Infections of the upper respiratory tract within 2 weeks prior to screening
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, lung function, or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study.
* HIV (Type I + Type II), hepatitis B or C, tuberculosis, or Sars-CoV-2 positive or not performed at visit 1
* Positive drug screen for methadone, cannabis, opiates, cocaine metabolites, amphetamines, barbiturates and benzodiazepines at visit 1
* History of drug or alcohol abuse
* Risk of non-compliance with study procedures
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study

COPD subjects

* Past or present disease other than COPD, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease or pulmonary disease (including but not confined to asthma, tuberculosis, bronchiectasis or cystic fibrosis).
* Regular intake of any prescribed or over the counter medication, which as judged by the investigator, may affect the outcome of the study or put the subject at risk because of participation in the study. Explicitly allowed is treatment with short-acting beta-2-agonists (SABA)/long-acting beta-2-agonists (LABA)/long-acting muscarinic-antagonists (LAMA), paracetamol for pain relief, oral contraceptive medication, hormonal replacement therapy, dietary and vitamin supplements. Not allowed are inhaled corticosteroids.
* Clinically relevant history of allergy as judged by the investigator.
* Intolerance against standard medication used during bronchoscopy, e.g. lidocaine, midazolam.
* Infections of the lower respiratory tract within 6 weeks prior to screening.
* Infections of the upper respiratory tract within 2 weeks prior to screening
* Exacerbation of COPD (treatment with oral or parenteral antibiotics and/or oral or parenteral glucocoterticosteroids (GCS) and/or hospitalization related to COPD) within 60 days of visit 1.
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, lung function, or ECG at Visit 1, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study.
* HIV (Type I + Type II), hepatitis B or C, tuberculosis, or Sars-CoV2 positive or not performed at visit 1.
* Positive drug screen for methadone, cannabis, opiates, cocaine metabolites, amphetamines, barbiturates and benzodiazepines at visit 1.
* History of drug or alcohol abuse.
* Risk of non-compliance with study procedures.
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Percentage of pH-Rhodo-positive alveolar macrophages | Ex-vivo, after collection of bronchoalveolar lavage (BAL) on Day 1
  Research compounds will be tested for the ability to influence the amount of efferocytosis against apoptotic cells, measuring the relative numbers of isolated alveolar macrophages that performed efferocytosis using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer ITEM Hannover, Germany
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No